CLINICAL TRIAL: NCT01851759
Title: A Random, Double-blind, Placebo- Controlled and Dose-finding, Multi-center, Phase II Clinical Trial of Methanesulfonic Acid Cinepazide Injection for Treatment of Acute Cerebral Infarction
Brief Title: Methanesulfonic Acid Cinepazide Injection for Treatment of Acute Cerebral Infarction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xijing005
Record Dates: First submitted 2013-05-07; First posted 2013-05-10 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — cinepazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cinepazide, Stroke, Injection (Experimental): Test drug：Methanesulfonic acid cinepazide injection（5ml/125mg）
  Interventions: Drug: cinepazide
- palcebo,Stroke,Injection (Placebo Comparator): Placebo：simulation agent of Methanesulfonic acid cinepazide injection（5ml sterile water for injection）
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cinepazide — 2 branches of Methanesulfonic acid cinepazide injection were matched into 250 ml 0.9% sodium chloride injection, iv gtt, speed is 100ml/h, once per day.
  1 branch of simulation agent of Methanesulfonic acid cinepazide injection was matched into 250 ml 0.9% sodium chloride injection, iv gtt, speed is 100ml/h, once per day.
  Other Names: Methanesulfonic acid cinepazide injection
  Arms: Cinepazide, Stroke, Injection
Drug: placebo — 2 branches of simulation agent of Methanesulfonic acid cinepazide injection were matched into 250 ml 0.9% sodium chloride injection, iv gtt, speed is 100ml/h, once per day.
  1 branch of simulation agent of Methanesulfonic acid cinepazide injection were matched into 250 ml 0.9% sodium chloride injection, iv gtt, speed is 100ml/h, once per day.
  Other Names: simulation agent of Methanesulfonic acid cinepazide
  Arms: palcebo,Stroke,Injection

SUMMARY:
Using placebo as control, The purpose of this study is to evaluate the efficacy and safety of methanesulfonic acid cinepazide injection to relieve disabled degree of acute cerebral infarction patients, and explore the best safe and effective dose as well as dose method.

DETAILED DESCRIPTION:
The study will enroll 288 acute cerebral infarction patients. Patients will be assigned randomly to receive either Methanesulfonic acid cinepazide injection or placebo treatment. All patient in the study will receive standard of care treatment and clinical, diagnostic, laboratory, safety, and follow-up evaluations. Follow-up evaluations, including National Institute of Health stroke scale(NIHSS), Barthel index score and modified Rankin scale assessments, will be done periodically until 90 days after onset. The degree of disabled improved will be a primary measure of drug effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 75 years old，male/ female；
2. The clinical diagnosis of first onset patients with anterior circulation infarction or who have suffered from stroke in history and complete recover from neurologic impairment (mRS score <2 before this disease）
3. Patients is proved by head skull CT and cerebral hemorrhage was excluded；
4. course of disease≤72h，the NIHSS score is ≥7 and ≤22；
5. Patients who voluntarily sign written informed consent. -

Exclusion Criteria:

1. Patients who suffer from cerebral infarction accompanied by disorder of consciousness, posterior circulation infarction, lacunar infarction and transient ischemic attack.
2. Patients who suffer from brain arteritis, brain tumor, brain injury, intracranial infection, brain parasitic disease, and so on . Patients who suffer from cardiac diseases such as rheumatic heart disease, coronary heart disease with atrial fibrillation .
3. Patients who suffer from severe complications, and expected survival period is within three months.
4. Patients require thrombolysis, anticoagulation, anti- fibrosis treatment .
5. Patients who suffer from serious brain artery stenosis that should go through interventional therapy .
6. Patients whose white blood cells or neutrophils is below the lower limit of the normal reference value .
7. Patients who have bleeding tendency or suffered from serious bleeding in 3 months.
8. Patients who have severe cardiac, liver and kidney disease, or whose kidney and liver function tests was abnormal（ALT,AST≥1.5 times of upper normal limit，Cr>upper normal limit）.
9. Patients who have complications of malignant tumor, serious or progressive disease in blood, digestion or other system.
10. Patients who have complications of mental illness un can not or do not want willing to cooperate .
11. Doubt or does have alcohol, drug abuse history
12. Allergic constitution or allergic to the test drug ingredients .
13. Pregnancy and lactation women or those who has a recent fertility plan
14. Patients who have participated in other clinical experiments three months before this test.
15. The patients who is unsuitable to participate in the clinical test in the view of researchers

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
modified Rankin scale | 3 month

SECONDARY OUTCOMES:
Barthel index | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, Doctor, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China